CLINICAL TRIAL: NCT07121322
Title: Phase II Study of Dornase Alfa and Cisplatin in Refractory Germ Cell Cancer.
Brief Title: Dornase Alfa and Cisplatin in Refractory Germ Cell Cancer.
Acronym: DACT-GCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT-SK-007
Record Dates: First submitted 2025-07-22; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Refractory Germ Cell Tumors; Dornase Alfa
Keywords: dornase alfa; refractory germ cell tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Non-randomized, open-label, single center trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dornase alfa and cisplatin (Experimental): Cisplatin 100mg/m2 day 1, every 3 weeks, Dornase alfa 125 microgram/kg day 1-5 i.v. push over 30 seconds±5 seconds
  Interventions: Drug: dornase alfa i.v. and cisplatin

INTERVENTIONS:
Drug: dornase alfa i.v. and cisplatin — Cisplatin 100mg/m2 day 1, every 3 weeks, Dornase alfa 125 microgram/kg day 1-5 i.v. push over 30 seconds±5 seconds

SUMMARY:
Germ cell tumors (GCTs) are highly curable malignancies; however, a subset of patients with relapsed or refractory disease after first- and second-line chemotherapy have a very poor prognosis, with long-term survival rates below 5%. New therapeutic strategies are needed in this setting. Emerging evidence indicates that extracellular DNA and markers of NETosis are associated with poor prognosis in GCTs, while DNase activity decreases with disease progression. Dornase alfa, a recombinant human DNase I approved for cystic fibrosis, may restore DNA homeostasis by degrading extracellular DNA. Preclinical studies demonstrated that dornase alfa, when combined with cisplatin, inhibited tumor growth in cisplatin-resistant GCT xenograft models. This proof-of-concept phase II study aims to evaluate the safety and efficacy of dornase alfa in combination with cisplatin in patients with relapsed or refractory GCTs, hypothesizing that extracellular DNA degradation by dornase alfa may enhance tumor control and restore cisplatin sensitivity.

DETAILED DESCRIPTION:
Germ cell tumors (GCTs) represent a unique solid tumor entity with high curability even in metastatic disease, primarily due to their marked chemosensitivity. Despite this, a subset of patients with multiple relapsed or refractory GCTs fail to achieve long-term remission with currently available standard- or high-dose salvage regimens. Long-term survival after failure of second-line chemotherapy is below 5%, underscoring the urgent need for new therapeutic strategies.

Recent translational research has highlighted a potential role of extracellular DNA and NETosis (neutrophil extracellular trap formation) in the pathogenesis and progression of refractory GCTs. Plasma analyses in GCT patients revealed elevated levels of cell-free DNA and NETosis markers in association with poor prognosis and disease burden. Moreover, reduced DNase activity during disease progression suggests impaired clearance of extracellular DNA, which may contribute to resistance to cytotoxic therapy.

Dornase alfa is a recombinant human deoxyribonuclease I (DNase I) approved for use in cystic fibrosis, where it enzymatically degrades extracellular DNA and reduces mucus viscosity. Preclinical in vitro experiments in TGCT cell lines, including cisplatin-resistant models, confirmed that dornase alfa is non-toxic at clinically relevant concentrations and does not negatively affect proliferation or migration. Notably, in vivo data from cisplatin-resistant xenograft models demonstrated that the combination of dornase alfa and cisplatin led to significant tumor growth inhibition, suggesting a potential synergistic effect mediated via degradation of extracellular DNA.

This is a non-randomized, open-label, single-center phase II study evaluating the efficacy and safety of dornase alfa in combination with cisplatin in adult male patients with histologically confirmed extracranial, metastatic, and multiply relapsed or refractory GCTs. The trial employs a Simon's optimal two-stage design.

The primary objective is to determine the 12-week progression-free survival (PFS) in the intent-to-treat population. Secondary objectives include overall response rate (ORR), PFS, overall survival (OS), safety, and the frequency of grade III/IV adverse events. An exploratory objective is to evaluate the association between clinical outcomes and circulating biomarkers (serum/plasma levels of DNase, cell-free DNA, and NETs).

Patients will receive intravenous cisplatin 100 mg/m² on day 1 of each 21-day cycle. Dornase alfa will be administered intravenously at a dose of 125 µg/kg daily on days 1-5. On day 1, dornase alfa will be given 2-3 hours after completion of cisplatin infusion; on subsequent days (2-5), it will be administered at the same time of day (±2 hours). Treatment will continue until disease progression or unacceptable toxicity.

Pharmacokinetic and biomarker studies will be conducted in each treatment cycle, with serum and plasma samples collected on day 1 and day 5 before administration of dornase alfa, and 4 and 24 hours post-administration. These will be used to monitor DNase activity, levels of cell-free DNA, and NETosis-related markers.

This study aims to provide proof-of-concept clinical evidence that targeting extracellular DNA with dornase alfa may enhance the anti-tumor efficacy of cisplatin in patients with heavily pretreated GCTs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Adult men aged 18 years or older.
3. ECOG (Eastern Cooperative Oncology Group) performance status: 0-1.
4. Histologically confirmed extracranial primary germ cell cancer, seminoma, or non-seminoma.
5. Rising serum markers (i.e., alfa-fetoprotein and human chorionic gonadotropin) on sequential measurement or biopsy-proven unresectable germ cell cancer.
6. Multiple relapsed/refractory GCTs (at least 2 lines of previous chemotherapy) and/or patients relapsing after high-dose chemotherapy or for patients non fit enough for high-dose chemotherapy.
7. Primary mediastinal GCTs in first relapse.
8. Patient's disease must not be amenable to cure with either surgery or chemotherapy in the opinion of investigator.
9. RECIST 1.1 measurable disease.
10. Adequate hematologic function defined by ANC > 1500/mm3, platelet count > 100 000/mm3 and hemoglobin level > 9g/dl.
11. Adequate liver function defined by a total bilirubin level < 1.5 ULN, and ALT, AST < 3 ULN or < 5 in case of liver metastases. For subjects with Gilbert's syndrome bilirubin > 1.5 × ULN is allowed if no symptoms of compromised liver function are present.
12. Adequate renal function: measured or calculated (by Cockcroft formula) creatinine clearance > 50 ml/min. Cockcroft formula: CLcr = [(140-age) x weight (Kg)]/[72 x creat (mg/dl)].
13. At least 4 weeks must have elapsed since the last radiotherapy and/or chemotherapy before study entry.
14. At least 4 weeks must have elapsed since the last major surgery.
15. Complete recovery from prior surgery, and/or reduction of all adverse events from previous systemic therapy or radiotherapy to grade 1.
16. Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
17. Male patients with a female partner of childbearing potential who agree to use an effective method of contraception (condom) and a highly effective method of contraception by their female partner during the study and 6 months after the last study treatment intake.

Exclusion Criteria:

1. Patients who do not fit inclusion criteria.
2. Other prior malignancy except successfully treated nonmelanoma skin cancer .
3. Other concurrent approved or investigational anticancer treatment, including surgery, radiotherapy, chemotherapy, biologic-response modifiers, hormone therapy, or immunotherapy.
4. Female patients.
5. Patients with other severe acute or chronic medical condition, or laboratory abnormality that would impair, in the judgment of investigator, excess risk associated with study treatment, or which, in judgment of the investigator, would make the patient inappropriate for entry into this study.
6. Hypersensitivity to any compound of the drugs, severe known allergies or intolerance to other recombinant protein products obtained from Chinese hamster ovary cells according to Investigatorś decision.
7. Known participation in another clinical trial investigating a drug and/or medical product in the last 30 days or 5 half-lives of the investigational drug and/or medicinal product (whichever is longer).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
12-week progresion-free survival | From enrollment to the end of treatment at 12 weeks
  12-week post-treatment initiation continuous progression-free survival rate will be summarized as counts and proportions with exact binomial 90% confidence interval (ITT population)

SECONDARY OUTCOMES:
Overall response rate | From the treatment initiation till the first response assessment at week 6
  Overall response rate (ORR) by RECIST 1.1 and tumor markers (AFP, HCG, LDH)
Progression-free survival | From the start of treatment (day 1) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  From the start of treatment (day 1) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Overall survival | Overall survival (OS) will be calculated from the start of treatment (day 1) until death from any cause assessed up to 100 months.
  Overall survival (OS) will be calculated from the start of treatment (day 1) until death from any cause assessed up to 100 months
Frequency of treatment related adverse events | From baseline through study completion, an average of 1 year
  Treatment related adverse reaction according to common toxicity criteria

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, prof., Study Chair — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
These data are confidential